CLINICAL TRIAL: NCT03411174
Title: Hypofractionated Partial Breast Irradiation After Breast-conserving Surgery for Low-risk Breast Cancer Patients
Brief Title: Hypofractionated PBI After BCS for Low-risk Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jinli Ma, Associate Professor of department of radiation oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-BC003
Record Dates: First submitted 2017-02-20; First posted 2018-01-26 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: breast cancer; hypofractionated partial breast irradiation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HF-PBI (Experimental): Hypofractionated partial breast irradiation was delivered to the tumor bed areas for low recurrence risk breast cancer patients, with prescription dose 40Gy in 15 fractions in 3 weeks.
  Interventions: Radiation: hypofractionated partial breast irradiation

INTERVENTIONS:
Radiation: hypofractionated partial breast irradiation — deliver 40Gy/15Fx to tumor bed areas

SUMMARY:
The study was designed to evaluate the feasibility and safety of hypofractionated partial breast irradiation after breast-conserving surgery for low-risk breast cancer patients.

DETAILED DESCRIPTION:
A total dose of 40.05Gy in 15 fractions was delivered to the tumor bed for each eligible breast cancer patients. The endpoints including loco-regional recurrence, cosmetic outcomes, and toxicities, were evaluated after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age≥ 50 years
* Treated with breast conversing surgery and sentinel lymph node biopsy or axillary lymph node dissection
* Negative surgical margins
* Pathologically confirmed invasive breast cancer
* A pathological T1N0M0 tumor -IHC: ER+/PR+/HER2-
* Tumor bed is labeled with Titanium clips
* Received adjuvant hormonal treatment
* No adjuvant chemotherapy
* ECOG:0-1
* Written informed consent.

Exclusion Criteria:

* Age<50 years
* KPS<70
* Treated with neoadjuvant chemotherapy
* Treated or being treated with chemotherapy
* With severe comorbidity
* Previous breast cancer or other malignant tumor history
* Previous radiotherapy for breast or thorax
* Medical contraindication for radiotherapy
* Pregnant or nursing

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2015-04; Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
The change of breast cosmetic outcome | Baseline, and three years after the completion of radiation therapy
  The breast cosmetic outcome was measured by Harvard 4 scale (poor, moderate, good, excellent) evaluation system

SECONDARY OUTCOMES:
Acute radiation-induced toxicity assessed by CTCAE v4.0 | 3weeks, 5weeks,1 and 3 months after treatment beginning
  acute toxicity related to skin and lung
Late complications | 3 years
  Complications related to radiation treatment after more than 3 months.
Ipsilateral breast tumor recurrence rate | 5 years
  The pathological confirmed tumor recurrence in the same breast
Local-regional recurrence | 5 years
  Disease recurrence in the ipsilateral chest wall or axillary, supraclavicular or infraclavicular fossa, or internal mammary chain.
Disease free survival | 5 years
  The interval from diagnosis to disease recurrence or death or last visit.
Overall survival | 5 years
  The interval from diagnosis to death or last visit

CONTACTS AND LOCATIONS:
Overall Officials: Jinli Ma, MD,PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang X, Wang X, Xu Z, Chu Y, Chen X, Zhang L, Meng J, Shi W, Yang Z, Mei X, Yu X, Zhang Z, Guo X, Mo M, Liu G, Wu J, Shao Z, Ma J. Hypofractionated partial breast irradiation after breast-conserving surgery for patients with early stage breast cancer in China Mainland: a single-arm prospective trial. Sci Rep. 2025 Jan 31;15(1):3869. doi: 10.1038/s41598-025-88600-5. PMID 39890895